CLINICAL TRIAL: NCT05476367
Title: Patients With Asymptomatic Hyperuricemia Have Stronger Local Inflammatory Response and Worse Outcome After Total Knee Arthroplasty
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Other Study IDs: 2021-0785
Record Dates: First submitted 2022-07-25; First posted 2022-07-27 (Actual); Last update posted 2022-07-27 (Actual); Status verified 2022-07

CONDITIONS: Arthritis Knee

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- patients with normal uric acid level: The uric acid level is below 420 μmol/L in men and 360 μmol/L in women
- patients with high uric acid level: The uric acid level is higher than 420 μmol/L in men and 360 μmol/L in women.

SUMMARY:
We identify all patients who had undergone primary total knee arthroplsty(TKA) from April 1, 2015, to March 30, 2016. Patients are grouped by uric acid level. The knee society score(KSS score) and the hospital for special surgery knee score (HSS score) before the surgery and 6 years after the surgery will be collected. Also the clinical data will be collected.

ELIGIBILITY:
Inclusion Criteria:

* patients who had undergone primary TKA from April 1, 2015, to March 30, 2016

Exclusion Criteria:

* (1) infection, (2) rheumatoid arthritis, (3) ankylosing spondylitis, (4) revision surgery, (5) patients with unicondylar knee replacement, (6) patients who have been diagnosed with gout or previous gouty symptoms, and (7) patients combined with preoperative redness or swelling.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All patients received primary TKA(totla knee arthroplasty) in our hospital.
Sampling Method: Probability Sample
Enrollment: 614 (Estimated)
Dates: Start 2022-08-01 (Estimated); Primary Completion 2022-09-01 (Estimated); Study Completion 2022-09-01 (Estimated)

PRIMARY OUTCOMES:
CRP | within 7 days after surgery
  C-reactive protein
temperature | within 7 days after surgery
  The nurses measured the body temperature by Non-contact Ear Thermometer. The temperatures were measured at 6 am, 14 pm, and 18 pm every day, and the patients were kept admitted till day 5. The highest one was chosen for analysis.
HSS score | 6 years after surgery
  the hospital for special surgery knee score
KSS scores | 6 years after surgery
  knee society score

REFERENCES:
- [Derived] Yu J, Mi T, Shao Z, Yan X. The Outcomes of Patients With Hyperuricemia After Total Knee Arthroplasty: A Retrospective Cohort Study. Orthop Surg. 2025 Dec;17(12):3477-3487. doi: 10.1111/os.70197. Epub 2025 Nov 6. PMID 41198532